CLINICAL TRIAL: NCT00727896
Title: "Reinforcement of Adherence to Prescription Recommendations in Diabetic Patients Using Short Message Service (SMS)- A Pilot Study"
Brief Title: "Information Technology Methodology for Patient Motivation in Diabetes Management."
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals (Other)
Responsible Party: Dr. Samith A Shetty/Consultant Diabetologist, INDIA DIABETES RESEARCH FOUNDATION (IDRF) and Dr. A. Ramachandran's Diabetes Hospitals (ARH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMS001IDRF
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-03

CONDITIONS: Type 2 Diabetes
Keywords: Life style modification,; Type 2 diabetes,; SMS,; Patient adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 is experimental with SMS (Experimental): Arm 1 is experimental with SMS intervention
  Interventions: Behavioral: Pre-coded messages
- 2 is (active comparator) standard care (Active Comparator): Arm 2 is the usual care arm (standard care)
  Interventions: Drug: Diabetes Treatment

INTERVENTIONS:
Behavioral: Pre-coded messages — Earlier life style modification and existing drug therapy was used and now SMS is added as a tool for reminder
  Arms: 1 is experimental with SMS
Drug: Diabetes Treatment — Life style modification and drug therapy
  Arms: 2 is (active comparator) standard care

SUMMARY:
Type 2 diabetes is a chronic metabolic disorder requiring lifestyle modification and medicines, adherence to which has to be practised on a daily basis.

Motivation of patients to adhere to treatment is difficult in clinical practice. It is well documented that majority of patients do not reach the glycaemic targets even in the centres of excellence. Regular short service messages (SMS) through cell phones could have a positive effect on behaviour and adherence to life style changes and compliance to drugs. It may be practical and feasible to use information technology as an effective and simple tool for motivating patients to adhere to the prescribed treatment regimen.

In diabetic patients, frequent reminders regarding the need for adherence to LSM and drugs by the medical professionals will improve the compliance.

DETAILED DESCRIPTION:
In diabetic patients, frequent reminders by the medical professionals on the need for adherence to Life Style Modification (LSM) and drugs will improve the compliance. SMS may be an effective and cheap tool of communication. Improved compliance is likely to result in better glycaemic control.

Out of total number of 200, consecutive randomization of 100 patients each to SMS or usual care arms will be done. Patients in the SMS group will get SMS once in 3 days as a reminder. Patients will be reviewed at 3, 6, 9 and 12 months from the date of randomization

Fasting and 2hr postprandial glucose and HbA1c will be tested during each visit.

At baseline and at the end of the study, lipids, and renal function test will also be done. A validated questionnaire will be used to assess physical activity, diet habits, adherence to drug prescriptions and frequency of monitoring of blood glucose. . Body weight, blood pressure, biochemical variables, scores for diet and physical activity and compliance to drugs, will be compared using students 't' test or chi-square test as relevant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 30-65 yrs of age at the time of entry and have type 2 diabetes for a minimum period of 5 years.
* HbA1C ranging 8.0-10.0%
* Patients either receiving OHA and / or insulin

Exclusion Criteria:

* Type 1 diabetes
* Patients with history of blindness, decreased vision
* Serious vascular complications :
* Cancer

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Behavioural changes resulting in diet, better adherence to treatment. | At intervals of three months for one year

SECONDARY OUTCOMES:
Reduction in HbA1c, other glycemic measures and improvement in blood lipid parameters | Annual

CONTACTS AND LOCATIONS:
Overall Officials: Samith A Shetty, M.B.B.S, MDRC, Principal Investigator — India Diabetes Research Foundation (IDRF) and Dr.A.Ramachandran's Diabetes Hospitals
Locations (1):
- India Diabetes Research Foundation and Dr.A.Ramachandran's Diabetes Hospitals, Chennai, Tamil Nadu, India

REFERENCES:
- [Background] Ramachandran A, Snehalatha C, Mary S, Mukesh B, Bhaskar AD, Vijay V; Indian Diabetes Prevention Programme (IDPP). The Indian Diabetes Prevention Programme shows that lifestyle modification and metformin prevent type 2 diabetes in Asian Indian subjects with impaired glucose tolerance (IDPP-1). Diabetologia. 2006 Feb;49(2):289-97. doi: 10.1007/s00125-005-0097-z. Epub 2006 Jan 4. PMID 16391903